CLINICAL TRIAL: NCT01911702
Title: MANAGEMENT OF THE PATIENT WITH ACUTE ABDOMEN SUBMITTED TO URGENT ABDOMINAL SURGERY: a Pilot Randomized Multicentre Study
Brief Title: Different Fluidic Strategy in Patients With Acute Abdomen : The Sure Volume
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Emanuela Biagioni, DR, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOModena
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Acute Abdomen
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Group (Active Comparator): In this group patients receive volemic standard treatment (conventional)
  Interventions: Other: Standard fluidic resuscitation.
- Restrictive Group (Active Comparator): In this group patients receive volemic small treatment (restrictive)
  Interventions: Other: Volemic small treatment

INTERVENTIONS:
Other: Standard fluidic resuscitation. — Goals:
  1. arterial pressure mean ≥ 65 mmHg or equal to the pre-operative
  2. diuretic rhythm ≥ 1 ml / Kg / h
  3. venous saturation in vena cava ≥ 70% or mixed venous saturation as Swan Ganz's catheter (SG) ≥ 65%
  4. BE> - 3
  5. Central Venous Pression (PVC) ≥ 8 mmHg; for patients undergoing mechanical ventilation, this limit may be raised to 12-15 mmHg.
  Arms: Conventional Group
Other: Volemic small treatment — Goals of the treatment:
  1. arterial pressure mean ≥ 60 mmHg or ≥ 10% less than the preoperative values
  2. diuretic rhythm ≥ 0.5 ml / kg / h
  3. venous saturation in vena cava ≥ 60% or mixed venous saturation ≥ 55% by SG
  4. BE> - 5
  5. PVC goal not necessary
  To achieve the therapeutic goals set out above will be executed a volemic fill up to values of PVC ≤ 5 mmHg or at maximum values of 2 mmHg more the incoming If after proper filling the targets aren't yet achieved, the patient will begin infusion of vasoactive drugs following the practice of department. If after 12 hours of admission the water balance will be > 10-15 ml / kg / h an infusion of furosemide should be initiated
  Arms: Restrictive Group

SUMMARY:
Acute abdomen is the clinical manifestation of irritation of the peritoneum, due to intra-abdominal generalized infection. With the exception of the primary ones which are the result of a bacterial translocation from the gastro-intestinal tract or an abdominal contamination for hematogenous way sometimes treatable with medical therapy alone, peritonitis represents a complex condition that requires an early surgical treatment.

Mortality linked to the peritonitis is extremely high and variable between 42% and 80% when associated with a systemic framework of severe sepsis. This variability is linked to a number of risk factors, including advanced age of the patients, the presence of comorbidity, male sex, a poor nutritional status, and a number of re-operations; as well as specific characteristics related to the type of infection, the timing of surgery, the beginning of an appropriate and early antibiotic therapy.The post-operative treatment of the patient with peritonitis significantly affects the outcome of the same. The presence of peritonitis and then the seizure of large volumes of liquids and the possible state of systemic vasodilation induced by the infectious process, provide a framework of hypovolemia. There is a literature that identifies in abdominal trauma damage patient's volemic aggressive resuscitation an element of pejorative outcomes. The purpose of this work is to evaluate the clinical changes determined by a different volemic strategy.

DETAILED DESCRIPTION:
DEPARTMENT OF GENERAL SURGERY AND SURGICAL SPECIALITIES SERVICE OF ANESTHESIOLOGY AND REANIMATION INTENSIVE CARE UNIT

Head: Prof. M. Girardis

MANAGEMENT OF THE PATIENT WITH ACUTE ABDOMEN SUBMITTED TO URGENT ABDOMINAL SURGERY: pilot study randomized multicentre

INTRODUCTION Acute abdomen is the clinical manifestation of irritation of the peritoneum, due to intra-abdominal generalized infection. Mortality linked to the peritonitis is extremely high and variable between 42% and 80% when associated with a systemic framework of severe sepsis. This variability is linked to a number of risk factors, including advanced age of the patients, the presence of comorbidity, male sex, a poor nutritional status, and a number of reoperations; as well as specific characteristics related to the type of infection, the timing of surgery, the beginning of an appropriate and early antibiotic therapy.

The post-operative treatment of the patient with peritonitis significantly affects the outcome of the same.

The centers involved in the study will be three:

1. post operative intensive care unit (ICU) - Modena University Hospital
2. reanimation unit - Carpi Hospital
3. intensive care unit (ICU) - Modena New Civil Hospital

OBJECTIVES PRIMARY OBJECTIVES: differences between the two treatment groups with different fluidic strategy in terms of 30-day mortality.

SECONDARY OBJECTIVES: differences between the two treatment groups with different fluidic strategy in terms of surgical complications, occurrence of organ failure, duration of mechanical ventilation and length of stay in ICU. Please refer to Section 6 for the definition of the endpoints / response variables for the secondary goals.

PLAN STUDY Study setting

The study will be conducted at the following facilities:

1. post operative intensive care unit (ICU) at Modena University Hospital
2. intensive care unit (ICU) at Modena Baggiovara
3. reanimation unit at Carpi Inclusion criteria All patients with acute abdomen undergoing abdominal surgery under emergency and presenting on arrival in ICU at least a sign of bad perfusion.

In the definition of acute abdomen, the following frameworks will be included:

1. primary peritonitis: bacterial contamination of the peritoneal cavity by microorganisms starting from extra-peritoneal sites (hematogenous in sepsis / bacteremia, from the female genital tract in the course of pelvic inflammatory disease (PID), from the retroperitoneum); translocation of microorganisms through the bowel
2. secondary peritonitis: bacterial contamination of the peritoneal cavity as a result of phlogosis or perforation of the digestive tract or female genital tract:

   1. acute abdominal infections (appendicitis, diverticulitis, cholecystitis, gallbladder empyema, suppurative cholangitis)
   2. other diseases (occlusion of the mesenteric, gastric or duodenal ulcer, strangulated hernia or volvulus, colic neoplasia, toxic megacolon, ruptured of intraperitoneal or visceral abscess)
   3. various intestinal diseases (tuberculosis, typhoid fever, cytomegalovirus (CMV) infection, infection with Clostridium)
   4. penetrating and not abdominal trauma (rupture or perforation of a hollow internal organ)
   5. surgical operation (stomach and duodenum, ileum, colon - rectum, bile - ducts) for dehiscence of anastomosis and / or sutures
3. tertiary or relapsing peritonitis, understood as persistent or recurrent peritonitis after apparently adequate medical and surgical treatment of secondary peritonitis
4. intestinal ischemia
5. pancreatitis with or without evidence of hemorrhagic- necrotic areas

The condition of hypoperfusion is identified by:

1. perioperative metabolic acidosis that can not be explained by other morbid conditions
2. arterial hypotension with PAM <60 mmHg or less than 15% of the preoperative

Exclusion Criteria

1. Patients with chronic renal failure already receiving dialysis treatment.
2. Acute Coronary Syndrome (ACS) <12 months and New York Hearth Classification (NHYA ) class > 3
3. Patients judged at the admission not subject to resuscitative measures for severity and comorbidity
4. Patients with massive hemorrhage in operative room or in the immediate perioperative with the need for blood transfusions and abundant blood products > 5 units of Erythrocyte Concentrates (EC)
5. Patients scheduled for Orthotopic Liver Transplantation (OLT)
6. Patients younger than 18 years old

In the definition of ACS, chest pain of suspected coronary origin with or without ST-segment elevation are included. According to the classification accepted by the European Society of Cardiology (ESC) and by the American College of Cardiology (ACC), the serum dosage of cardiac troponins can make the diagnosis of myocardial infarction.

STUDY PROCEDURES Screening and inclusion

At the entrance to the ICU all patients that meet the criteria for inclusion and don't present exclusion criteria - will be evaluated for randomization.

The attending physician will have to notify the coordinating center as soon deemed to have identified a patient to be enrolled. The coordinating center is at the Intensive Care Unit of the University Hospital of Modena.

Randomization must be done at the time of admission to ICU.

The method of randomization will be by "parallel group", the type of simple randomization and the randomization list will be obtained through the use of a random number generator computerized in a 1:1 ratio. Patients who meet the inclusion criteria are assigned over the telephone by medical coordinator:

1. or to the group receiving volemic standard treatment (conventional)
2. or to the group receiving volemic small treatment (restrictive) The contact number for randomization is always 0594224896

Group "conventional"

Goals of the treatment:

1. arterial pressure mean ≥ 65 mmHg or equal to the pre-operative
2. diuretic rhythm ≥ 1 ml / Kg / h
3. venous saturation in vena cava ≥ 70% or mixed venous saturation as Swan Ganz's catheter (SG) ≥ 65%
4. base excess (BE) > - 3
5. Central Venous Pression (PVC) ≥ 8 mmHg; for patients undergoing mechanical ventilation, this limit may be raised to 12-15 mmHg.

To achieve the therapeutic goals set out above will be executed a volemic fill until reaching central venous pressure values of 8-10 mmHg. Crystalloid solutions and specifically balanced III, Ringer solutions or alternatively glucose solution will be infused at 5% in patients with serum sodium ≥ 145 milliequivalent (mEq) / L.

For this group of patients, the overall water balance won't be binding. If after proper filling the targets aren't yet achieved, the patient will begin infusion of vasoactive drugs following the practice of department.

If you are unable to get a goal value of venous saturation you can consider:

1. The chance to infuse additional volumes of fluids
2. the chance to transfuse concentrate red blood cells
3. The chance to infuse dobutamine up to 20 microg / kg / min

Group "restrictive"

Goals of the treatment:

1. arterial pressure mean ≥ 60 mmHg or ≥ 10% less than the preoperative values
2. diuretic rhythm ≥ 0.5 ml / kg / h
3. venous saturation in vena cava ≥ 60% or mixed venous saturation ≥ 55% by SG
4. BE> - 5
5. PVC goal not necessary

To achieve the therapeutic goals set out above will be executed a volemic fill up to values of PVC ≤ 5 mmHg or at maximum values of 2 mmHg more the incoming If after proper filling the targets aren't yet achieved, the patient will begin infusion of vasoactive drugs following the practice of department. If after 12 hours of admission the water balance will be > 10-15 ml / kg / h an infusion of furosemide should be initiated in order to bring the budget of the patient to 10-15 ml / kg in 24 hours.

DATA COLLECTION Data Collection Program

Data collection will be done by compiling data collection forms. In particular, the following types of data collection formats will be filled:

1. basal and randomization card (Record Form 1)
2. card to 6 hours after randomization (Record Form 2)
3. 24 hours card (Record Form 3)
4. daily continuation card (as long as the patient is admitted to Post Operative Intensive Therapy, Record Form 4)
5. Conclusion card (Record Form 5)

The basal card will contain:

1. patient's personal details
2. information according with remote and proximal medical history
3. patient's vital parameters
4. patient's therapy

The final board will collect data until it will be verified:

1. patient's discharge from the hospital
2. thirtieth day of hospitalization
3. patient's death

END POINT / VARIABLE RESPONSE

Study end point:

1. Primary: Mortality at 30 days
2. Secondary:

   1. Number of surgical complications (anastomotic dehiscences, need for re-operation, need for percutaneous drainages of evacuation, the development of abdominal hypertension).
   2. Occurrence of acute respiratory failure identified with respiratory exchanges with values of P / F less than 300 mmHg
   3. Occurrence of lack of circulation with the use of vasoactive amines in the post-operative
   4. Occurrence of acute renal failure (number of extracorporeal treatments and / or serum creatinine ≥ 1.9 mg / dl)
   5. Occurrence of hepatic insufficiency with serum total bilirubin values greater than 2.0 mg / dl
   6. Days of mechanical ventilation
   7. Days of ICU staying

In the definition of surgical complications all the following situations are included:

1. anastomotic dehiscences
2. the need for reoperation
3. the need to place percutaneous drainages of evacuation
4. wound infection that requires surgical toilet or with microbiological samples positive

The accepted definition of abdominal hypertension is hypertension of the abdominal cavity of retroperitoneal, intraperitoneal or parietal origin. The measurement system accepted in the study is exclusively that one of the intravesical bladder catheterization. The values considered as reference are:

1. mild abdominal hypertension: 10-20 mmHg
2. moderate abdominal hypertension: 20-40 mmHg
3. severe abdominal hypertension: > 40 mmHg The numeric variables which indicate organ failure shall be guided by the SOFA score for severity score ≥ 2. In extracorporeal treatments hemo-filtration sessions with both intermittent and continuous methods are considered.

SIZE OF THE STUDY AND DATA ANALYSIS CRITERIA This is a phase II study, which is exploratory and estimative and that involves randomization of all recruitable patients during the period of study all over the three centers involved in the work. The study will begin on January 2010 and will last for 3 years. The sample size has been calculated on the basis of the available data at the Post-Operative Intensive Care Unit of the Hospital in 2007: these data showed a mortality of the patients with acute abdomen undergoing abdominal surgery under emergency and presenting at the moment of arrival to Post Operative Intensive Therapy at least a sign of hypoperfusion of 30%. Assuming a two-tailed alpha level <0.05 and a power of 80%, we have calculated that 100 patients per arm are needed to detect an absolute reduction in mortality of 15%. This reduction appears to be significant from the clinical point of view considering previous trials of fluidic therapy in shocked patients . For comparisons between the means, the t-student test will be used. For comparison of events frequencies the χ2 test or Fisher's test - as indicated - will be used. A p <0.05 will be considered statistically significant. Static analysis will be performed using version 16.0 of SPSS software.

ELIGIBILITY:
Inclusion Criteria:

All patients with acute abdomen undergoing abdominal surgery under emergency and presenting on arrival in ICU at least a sign of bad perfusion.

Exclusion Criteria:

1. Patients with chronic renal failure already receiving dialysis treatment
2. Acute Coronary Syndrome (ACS) <12 months and New York Hearth Classification (NHYA ) class > 3
3. Patients judged at the admission not subject to resuscitative measures for severity and comorbidity
4. Patients with massive hemorrhage in operative room or in the immediate perioperative with the need for blood transfusions and abundant blood products > 5 units of Erytrocyte Concentrates (EC)
5. Patients scheduled for Orthotopic Liver Transplantation (OLT)
6. Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
differences between the two treatment groups with different fluidic strategy in terms of 30-day mortality. | within the first 30 days after surgery
  The purpose of this work is to evaluate the clinical changes determined by a different volemic strategy.

SECONDARY OUTCOMES:
differences between the two treatment groups with different fluidic strategy in terms of surgical complications | within the forst 30 days after surgery
differences between the two treatment groups with different fluidic strategy in terms of occurrence of organ failure, | within the first 30 days after surgery
differences between the two treatment groups with different fluidic strategy in terms of duration of mechanical ventilation | within the first 30 days after surgery
differences between the two treatment groups with different fluidic strategy in terms of length of stay in ICU | within 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Girardis, Professor, Study Chair — Azienda Ospedalier Universitaria di Modena

REFERENCES:
- [Background] Streat SJ, Plank LD, Hill GL. Overview of modern management of patients with critical injury and severe sepsis. World J Surg. 2000 Jun;24(6):655-63. doi: 10.1007/s002689910107. PMID 10773117
- [Background] Raymond DP, Pelletier SJ, Crabtree TD, Schulman AM, Pruett TL, Sawyer RG. Surgical infection and the aging population. Am Surg. 2001 Sep;67(9):827-32; discussion 832-3. PMID 11565758
- [Background] Farinas-Alvarez C, Farinas MC, Fernandez-Mazarrasa C, Llorca J, Casanova D, Delgado-Rodriguez M. Analysis of risk factors for nosocomial sepsis in surgical patients. Br J Surg. 2000 Aug;87(8):1076-81. doi: 10.1046/j.1365-2168.2000.01466.x. PMID 10931054
- [Background] Stafford RE, Weigelt JA. Surgical infections in the critically ill. Curr Opin Crit Care. 2002 Oct;8(5):449-52. doi: 10.1097/00075198-200210000-00013. PMID 12357114
- [Background] Madigan MC, Kemp CD, Johnson JC, Cotton BA. Secondary abdominal compartment syndrome after severe extremity injury: are early, aggressive fluid resuscitation strategies to blame? J Trauma. 2008 Feb;64(2):280-5. doi: 10.1097/TA.0b013e3181622bb6. PMID 18301187
- [Background] Cotton BA, Guy JS, Morris JA Jr, Abumrad NN. The cellular, metabolic, and systemic consequences of aggressive fluid resuscitation strategies. Shock. 2006 Aug;26(2):115-21. doi: 10.1097/01.shk.0000209564.84822.f2. PMID 16878017
- [Background] Marshall JC, Innes M. Intensive care unit management of intra-abdominal infection. Crit Care Med. 2003 Aug;31(8):2228-37. doi: 10.1097/01.CCM.0000087326.59341.51. PMID 12973184
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437